CLINICAL TRIAL: NCT03647527
Title: Predictive Factor Analysis of Acute Radiation Oral Mucositis in Nasopharyngeal Carcinoma Patients Treated With Precise Radiotherapy Technique Combined Chemotherapy
Brief Title: Predictor Analysis of Acute Radiation Oral Mucositis in NPC Patients Treated With IMRT/TOMO Combined Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen yuanyuan, Clinical Professor, Zhejiang Cancer Hospital
Other Study IDs: PF-AROM-NPC-IMRT/TOMO
Record Dates: First submitted 2018-08-09; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; acute radiation oral mucositis; intensity modulated radiotherapy; tomography radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiation induced oral mucositis which may result in reduced quality of life is commonly seen during radiotherapy, especially combined with chemotherapy. This study is a prospective, single center, and exploratory study. Two contour methods of oral mucosal will be used in this study. All detail information will be recorded prospectively. The aim of this study is to explore predictive factors of acute radiotherapy induced oral mucositis in nasopharyngeal carcinoma patients treated with new precise radiotherapy (intensity modulated radiotherapy or tomography radiotherapy) by using different dosimetric parameters and clinically relevant variables.

DETAILED DESCRIPTION:
To prospectively identify the predictive value of different dosimetric parameters and assess the predictors of acute radiation oral mucositis in nasopharyngeal carcinoma patients treated with intensity modulated radiotherapy or tomography radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1.Clinical diagnosis of nasopharyngeal carcinoma. 2.7th version American Joint Committee on Cancer (AJCC) stage II-IVB. 3.Age must above 18. 4.Performance status must be 0 or 1 according to Eastern Cooperative Oncology Group.

5.Adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

1. Treatment with palliative intent.
2. Previous malignancy.
3. Pregnancy or lactation.
4. A history of previous radiotherapy, chemotherapy, or surgery (except diagnostic) to the primary tumor or nodes.
5. Any severe coexisting disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between September 2016 and August 2018, consecutive patients with II-IVB nasopharyngeal carcinoma receiving intensity modulated radiotherapy or tomography radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
the highest grade of oral mucositis | oral mucocitis will be checked every day during the date of initiation of radiation therapy until the date of completion of radiation therapy, the highest grade ≥ 3 define as severe oral mubocitis, assessed up to a month and a half
  Radiation Therapy Oncology Group/European Organization for research and treatment acute radiation morbidity scoring criteria. Grade 0: No change over baseline, Grade 1: Injection/ may experience mild pain not requiring analgesic, Grade 2: Patchy mucositis which may produce an inflammatory serosanguinitis discharge/ may experience moderate pain requiring analgesia, Grade 3: Confluent fibrinous mucositis/ may include severe pain requiring narcotic, Grade 4: Ulceration, hemorrhage or necrosis, Grade 5: death (Higher score equals to worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Chen, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No